CLINICAL TRIAL: NCT03000400
Title: The Family as a Resource for Improving Patient and Family Functioning After Traumatic Brain Injury. A Randomized Controlled Trial of a Family Centered Intervention
Brief Title: Family Centered Intervention After Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Extra Foundation for Health and Rehabilitation (Other); The National Association for the Traumatically Injured, Norway (Unknown); Baerum municipality, Department of Rehablitation, Norway (Unknown)
Responsible Party: Principal Investigator, Helene Lundgaard Søberg, Senior researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/1215/REK sør-øst C
Record Dates: First submitted 2016-11-11; First posted 2016-12-22 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Patient and family members receiving the 8 week family centered intervention, The Traumatic Brain Injury Family System Intervention.
  Interventions: Behavioral: The Traumatic Brain Injury Family System Intervention.
- Control group (Active Comparator): Family members attend one ongoing psycho-educational group session provided by Oslo University Hospital (OUH).
  Interventions: Behavioral: Psycho-educational session at OUH

INTERVENTIONS:
Behavioral: The Traumatic Brain Injury Family System Intervention. — Theoretically based intervention consisting of 8 weekly 90 minutes sessions addressing specific topics according to a manual.
  Arms: Intervention group
Behavioral: Psycho-educational session at OUH — 2.5 hour psycho-educational session for the patient's family members.
  Arms: Control group

SUMMARY:
The purpose of this study is to determine the effectiveness of a multi-professional theoretically based family centered intervention, The Traumatic Brain Injury Family System Intervention (TBIFSI), for the family members and TBI patients in improving family dynamics and functioning. The intervention will be provided in collaboration with the municipal rehabilitation service. The intervention group will be compared with a control group receiving treatment as usual, defined as an individually tailored multidisciplinary approach, and the family members will attend one ongoing psycho-educational group session of 2.5 hour provided by Oslo University Hospital (OUH).

ELIGIBILITY:
Inclusion Criteria:

Patients: Home dwelling individuals age 16-65 who have sustained a TBI and receiving health services. They should:

1. Be out of post traumatic amnesia for at least one month
2. Have been discharged from post-acute rehabilitation in the specialized health care system in the last 6 - 18 months
3. Have a Ranchos Los Amigos Scale score of at least 8
4. Mini Mental Status Examination score >23

   * Family members: individuals related by blood or marriage/cohabitating with the TBI patient.

     1. Belongs to the same household as the individual with TBI and/or in close relation with the patient
     2. are between 18-65 years of age.

Exclusion Criteria:

* TBI survivors or their family members with a history of psychiatric or neurologic illness, active learning disability, or active substance abuse. Inability to speak and read Norwegian. Families in which there are other members requiring care or who have previously been caregivers for other family members.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Change in Short Form 36 Health Survey (SF-36) Mental Component Summary | Baseline at study start, at 8 weeks after inclusion, 6 months after completion of the intervention
  Mental health for all study participants
Change in Caregiver Burden Scale (CBS) | Baseline at study start, at 8 weeks after inclusion, 6 months after completion of the intervention
  Caregiver Burden for the family members

SECONDARY OUTCOMES:
Quality of Life after Traumatic Brain Injury (QOLIBRI) | Baseline at study start, at 8 weeks after inclusion, 6 months after completion of the intervention
  Quality of Life for the patients
Faces IV | Baseline at study start, at 8 weeks after inclusion, 6 months after completion of the intervention
  Family dynamics for all study participants

OTHER OUTCOMES:
Resilience Scale for Adults (RSA) | Baseline at study start, at 8 weeks after inclusion, 6 months after completion of the intervention
  Resilience for all study participants
The Generalized Self-Efficacy Scale | Baseline at study start, at 8 weeks after inclusion, 6 months after completion of the intervention
  Self-efficacy for all participants
The TBI Self-Efficacy Scale | Baseline at study start, at 8 weeks after inclusion, 6 months after completion of the intervention
  Self-efficacy for the patients
Patient Health Questionnaire 9 (PHQ-9) | Baseline at study start, at 8 weeks after inclusion, 6 months after completion of the intervention
  Mental health for all participants
The Generalized Anxiety Disorder 7 (GAD-7) | Baseline at study start, at 8 weeks after inclusion, 6 months after completion of the intervention
  Mental health for all participants

CONTACTS AND LOCATIONS:
Overall Officials: Helene L. Soberg, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway